CLINICAL TRIAL: NCT06356649
Title: Investigation of the Effects of Pressure Support Ventilation and Positive Airway Pressure Modes on Respiratory System Complications During Extubation
Brief Title: Investigation of the Effects of Pressure Support Ventilation and Positive Airway Pressure Modes During Extubation
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Dilek Cetinkaya, Associate Professor, Eskisehir Osmangazi University
Other Study IDs: ESOGU2
Record Dates: First submitted 2024-03-31; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia
Keywords: pressure controlled ventilation; positive end-expiratory pressure; tracheal extubation
MeSH Terms: interventions — Airway Extubation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Goup 1: Patients extubated after general anesthesia
  Interventions: Procedure: extubation
- Group 2: Patients with complications after extubation
  Interventions: Procedure: extubation

INTERVENTIONS:
Procedure: extubation — Complications after extubation

SUMMARY:
Controlled ventilation is applied to patients intubated for general anesthesia. Additionally, positive end-expiratory pressure (PEEP) and pressure support are mechanical ventilation modes that have been used in general anesthesia practice for many years. When the recovery-extubation phase is reached, intermittent bag-mask ventilation is usually used and the patient is allowed to breathe spontaneously and is extubated when an adequate respiratory level is reached. It has been shown in previous studies that the use of intermittent mask ventilation causes postoperative atelectasis. Different methods have been used to prevent postoperative atelectasis. In our study, we aimed to observe the effect of terminating general anesthesia at the end of the operation and using PEEP and pressure-supported ventilation during the extubation phase on early complications.

DETAILED DESCRIPTION:
After informed consent was obtained from the patients, monitoring was performed as we practice in routine anesthesia practice. Pressure controlled ventilation (PCV) mode and positive end-expiratory pressure (PEEP) were used as the mechanical ventilation mode after intubation. After the operation was completed, PCV mode on the mechanical ventilator was continued until the patient was extubated. Afterwards, patients were extubated if they complied with verbal commands and/or swallowed and/or coughed in response to vocal stimuli, pupils were in the midline and conjugated, BIS value was >80, breathing was regular, and TOF response was >90%. Hemodynamic and respiratory system complications were recorded during the intraoperative, recovery-extubation and postoperative periods. Patients over the age of 18 with American Society of Anesthesiology physical classification (ASA) 1-3 who underwent laparoscopic cholecystectomy were included in the study. In the preoperative period, the patient's demographic data and hemodynamic data, and in the intraoperative period, respiratory data (tidal volume, pressure applied during inspiration, peep, etc.) and hemodynamic data were recorded. Complications recorded during recovery-extubation; desaturation, laryngospasm, bronchospasm, agitation, rescue mask ventilation application, airway obstruction, nausea-vomiting, re-intubation, struggling.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 with American Society of Anesthesiology physical classification (ASA) 1-3 who underwent laparoscopic cholecystectomy were included in the study

Exclusion Criteria:

* The patient does not want to participate in the study.
* Known advanced lung disease, advanced-stage heart disease
* Switching from laparoscopic surgery to open surgery
* Surgical procedure exceeds 120 minutes
* intraoperative bleeding >500 ml

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing laparoscopic anesthesia with general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Complications developing during recovery-extubation | 1 hour
  desaturation, laryngospasm, bronchospasm, agitation, rescue mask ventilation application, airway obstruction, nausea-vomiting, re-intubation, struggling.

SECONDARY OUTCOMES:
hemodynamic changes | first 24 hours
  heart rate
hemodynamic data | during 24 hours
  mean arterial pressure

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Çetinkaya, Principal Investigator — Eskisehir Osmangazi University
Locations (1):
- Eskisehir Osmangazi University Medical Faculty, Eskişehir, Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel RI, Hannallah RS, Norden J, Casey WF, Verghese ST. Emergence airway complications in children: a comparison of tracheal extubation in awake and deeply anesthetized patients. Anesth Analg. 1991 Sep;73(3):266-70. PMID 1867418
- [Background] Jeong H, Tanatporn P, Ahn HJ, Yang M, Kim JA, Yeo H, Kim W. Pressure Support versus Spontaneous Ventilation during Anesthetic Emergence-Effect on Postoperative Atelectasis: A Randomized Controlled Trial. Anesthesiology. 2021 Dec 1;135(6):1004-1014. doi: 10.1097/ALN.0000000000003997. PMID 34610099
- [Result] Juang J, Cordoba M, Ciaramella A, Xiao M, Goldfarb J, Bayter JE, Macias AA. Incidence of airway complications associated with deep extubation in adults. BMC Anesthesiol. 2020 Oct 29;20(1):274. doi: 10.1186/s12871-020-01191-8. PMID 33121440
- [Derived] Ata AR, Cetinkaya D, Yaman F. Investigating the effects of pressure support ventilation and positive end-expiratory pressure during extubation on respiratory system complications. Perioper Med (Lond). 2024 Dec 18;13(1):118. doi: 10.1186/s13741-024-00477-6. PMID 39696646